CLINICAL TRIAL: NCT03839940
Title: Phase III Placebo-Controlled Trial to Evaluate Dexamethasone Use for Everolimus-Induced Oral Stomatitis: Prevention Versus Early Treatment Approaches: MIST (My Individualized Stomatitis Treatment)
Brief Title: Dexamethasone in Reducing Everolimus-Induced Oral Stomatitis in Patients With Cancer
Acronym: MIST
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Severe lack of accrual
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: A221701; NCI-2018-02648 (Registry Identifier: NCI Clinical Trial Reporting Program); UG1CA189823 (NIH)
Record Dates: First submitted 2019-02-06; First posted 2019-02-15 (Actual); Results first posted 2022-08-01 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Dexamethasone; Surveys and Questionnaires; Everolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (dexamethasone) (Experimental): Patients receive 10mg oral everolimus daily as standard of care and 10ml dexamethasone oral mouthwash, swished for 2-minutes daily, for 8 weeks.
  Interventions: Drug: Dexamethasone; Other: Questionnaire; Other: Quality-of-Life Assessment; Drug: Everolimus
- Group II (placebo) (Placebo Comparator): Patients receive 10mg oral everolimus daily as standard of care and 10ml placebo oral mouthwash, swished for 2-minutes daily, for 8 weeks.
  Interventions: Other: Placebo; Other: Questionnaire; Other: Quality-of-Life Assessment; Drug: Everolimus

INTERVENTIONS:
Drug: Dexamethasone — Given as mouthwash
  Arms: Group I (dexamethasone)
Other: Placebo — Given as mouthwash
  Arms: Group II (placebo)
Other: Questionnaire — Ancillary studies
Other: Quality-of-Life Assessment — Ancillary studies
Drug: Everolimus — Standard of care

SUMMARY:
This phase III trial studies how well dexamethasone works in reducing everolimus-induced oral stomatitis in patients with cancer. Dexamethasone may help to reduce the everolimus-induced oral stomatitis so as to improve quality of life in cancer patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if the initiation of dexamethasone at the start of everolimus treatment prevents mTOR inhibitor-associated stomatitis (mIAS)-associated pain, compared to the initiation of placebo.

II. To determine if the initiation of dexamethasone at the start of everolimus treatment will be superior compared to the initiation of placebo in terms of the overall severity of mIAS-associated pain.

SECONDARY OBJECTIVES:

I. To utilize the same measurement method that was reported in the SWISH trial: A combination of a patient reported pain scale, data from a normalcy of diet questionnaire, and clinician grading of stomatitis to determine the incidence of > grade 2 mIAS.

II. To determine if the initiation of dexamethasone at the start of everolimus increases time to development of mouth pain using daily numerical analog scale patient-reported data collection.

III. To assess if quality of life is better when dexamethasone mouth rinse use starts at the same time as everolimus use versus at the time when mouth pain begins.

IV. To investigate if starting dexamethasone mouth rinse concurrent with starting everolimus improves patients' ability to adhere to everolimus therapy.

V. To compare dexamethasone prescription fill rates and timing between patients who received placebo versus study drug at the initiation of everolimus.

Trial Design:

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive everolimus orally (PO) once daily (QD) as standard of care and dexamethasone as mouthwash over 2 minutes 4 times per day (QID) for 8 weeks.

GROUP II: Patients receive everolimus PO QD as standard of care and placebo as mouthwash over 2 minutes QID for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Current cancer diagnosis, about to receive oral everolimus 10 mg/day with or without an endocrine agent. Patients about to receive everolimus for off label use for any cancer are also eligible.
* Not currently receiving chemotherapy or any other agent known to cause mucositis or stomatitis. Trastuzumab and ovarian function suppression are allowed.
* Any prior chemotherapy or other stomatitis/mucositis-causing therapy must be completed at least 2 weeks prior to registration.
* Not currently suffering from stomatitis/mucositis or mouth ulcers. Patients should not have had any stomatitis or mouth pain for at least 7 days prior to registration.
* Patients should not receive any other agent which would be considered treatment for stomatitis or impact the primary endpoint.
* No history of candida infection (thrush) within the last 3 months.
* Not currently being treated with corticosteroids.
* No uncontrolled diabetes mellitus, defined by hemoglobin A1C greater than 8%, although A1C is not needed for all patients, hemoglobin (Hgb)A1C < 8 is required for everyone with diabetes or suspected diabetes.
* Patients must be able to read and comprehend English. Local translation, including verbal translation of professionals (PROs) is not permitted.
* Not pregnant and not nursing, because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown. Therefore, for women of childbearing potential only, a negative pregnancy test done =< 7 days prior to registration is required.
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2021-01-08 (Actual); Study Completion 2022-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Ruddy, MD, Study Chair — Mayo Clinic
Locations (319):
- United States (319):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Kingman Regional Medical Center, Kingman, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - PCR Oncology, Arroyo Grande, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Trinity Regional Medical Center, Fort Dodge, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Ochsner LSU Health Monroe Medical Center, Monroe, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Mercy Medical Center, Springfield, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - IHA Hematology Oncology Consultants-Brighton, Brighton, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - IHA Hematology Oncology Consultants-Canton, Canton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - IHA Hematology Oncology Consultants-Chelsea, Chelsea, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China Township, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Academic Hematology Oncology Specialists, Grosse Pointe Woods, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Huron Medical Center PC, Port Huron, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Great Lakes Cancer Management Specialists-Rochester Hills, Rochester Hills, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Ascension Saint Joseph Hospital, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - IHA Hematology Oncology Consultants-Ann Arbor, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Southeast Nebraska Cancer Center - 68th Street Place, Lincoln, Nebraska
  - Faith Regional Health Services Carson Cancer Center, Norfolk, Nebraska
  - Great Plains Health Callahan Cancer Center, North Platte, Nebraska
  - Nebraska Cancer Specialists - Omaha, Omaha, Nebraska
  - Oncology Hematology West PC, Omaha, Nebraska
  - Regional West Medical Center Cancer Center, Scottsbluff, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - 21st Century Oncology-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Oakey, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - 21st Century Oncology-Vegas Tenaya, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology-Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Virtua Samson Cancer Center, Moorestown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Hematology Oncology Associates of Central New York-Auburn, Auburn, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Hematology Oncology Associates of Central New York-Onondaga Hill, Syracuse, New York
  - CaroMont Regional Medical Center, Gastonia, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Southpointe-Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Central Ohio Breast and Endocrine Surgery, Gahanna, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Self Regional Healthcare, Greenwood, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Overlake Medical Center, Bellevue, Washington
  - Valley Medical Center, Renton, Washington
  - Legacy Cancer Institute Medical Oncology and Day Treatment, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Mayo Clinic Health System Eau Claire Hospital-Luther Campus, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - Marshfield Clinic - Ladysmith Center, Ladysmith, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

IPD SHARING:
Plan to Share IPD: Yes
Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive
URL: https://nctn-data-archive.nci.nih.gov/

REFERENCES:
- [Derived] Ruddy KJ, Zahrieh D, He J, Waechter B, Holleran JL, Lewis LD, Chow S, Beumer J, Weiss M, Trikalinos N, Faller B, Lustberg M, Rugo HS, Loprinzi C. Dexamethasone to prevent everolimus-induced stomatitis (Alliance MIST Trial: A221701). Semin Oncol. 2023 Feb-Apr;50(1-2):7-10. doi: 10.1053/j.seminoncol.2023.01.001. Epub 2023 Jan 17. PMID 36693773
- Available data/document: Individual Participant Data Set — https://nctn-data-archive.nci.nih.gov/ — Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group I (Dexamethasone) | Group II (Placebo)
Started | 20 | 19
Completed | 16 | 17
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — No Post-Baseline Pain Score Data | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I (Dexamethasone) | Group II (Placebo) | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (10.71) | 65.3 (8.46) | 65.3 (9.46)
Age, Customized [Count of Participants; unit: Participants]
  Age group: <50 years | 1 | 1 | 2
  Age group: 50 - 65 years | 8 | 7 | 15
  Age group: >65 years | 7 | 9 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 16 | 31
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 12 | 16 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Cancer Type [Count of Participants; unit: Participants]
  Breast | 11 | 12 | 23
  Other | 5 | 5 | 10
ECOG Performance Status [Count of Participants; unit: Participants] — ECOG = 0: Fully active, able to carry on all pre-disease performance without restriction.
  ECOG = 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  ECOG = 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours.
  ECOG = 0 is better. ECOG = 2 is worse.
  Participants
    0 | 8 | 7 | 15
    1 | 7 | 10 | 17
    2 | 1 | 0 | 1
Continuous Patient Reported Mouth-Pain Score [Mean (Standard Deviation); unit: scores on a scale] — Pain scale from 1-10. 1 is better and 10 is worse.
  scores on a scale | 0 (0) | 0.1 (0.24) | 0.03 (0.17)
Discrete Patient Reported Mouth-Pain Score [Count of Participants; unit: Participants] — Mouth-Pain score = 0: Patient has no pain in their mouth. Mouth-Pain score > 0: Patient has pain in their mouth. Mouth-Pain score = 0 is better. Mouth-Pain score > 0 is worse.
  Participants
    = 0 | 16 | 16 | 32
    > 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of the mTOR Inhibitor-associated Stomatitis (mIAS)-Related Pain Based on Daily Self-reports Via the Numerical Analogue Scale
Description: The numerical analogue mouth pain score (NAMPS) is a single item measured on a 0 to 10 scale, with 0 corresponding to "No pain" and 10 corresponding to "Pain as bad as it can be." Will compare the incidence rate of any mouth pain (i.e., any score greater than 0) as assessed by the NAMPS between the prevention versus early treatment approaches using a Chi-square test.
Time Frame: Up to 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Dexamethasone) | Group II (Placebo)
Number analyzed (Participants) | 16 | 17
Participants
  No Pain | 7 | 8
  Pain | 9 | 9
Statistical Analysis 1: Comparison: Group I (Dexamethasone) vs Group II (Placebo); Test type: Superiority; p < 0.9999, Fisher Exact

2. Primary Outcome: Severity of Mouth Pain Scores
Description: Average Area Under the Curve per assessment (aAUCpa) of mouth pain scores as measured by NAMPS will be computed for each patient to summarize the sequence of numerical analogue mouth pain scores over the eight week study period. Scores are reported on a 0-100 scale, where 100 = better outcome QOL (i.e. less pain). The aAUCpa is the average of each AUC between each sequential assessment from treatment-initiation to the end of the treatment at 8 weeks post-treatment-initiation and will be compared between the two treatment arms.
Time Frame: Up to 8 weeks
Measure: Mean (Standard Deviation); unit: scores on scale * days
Groups:
- Group I (Dexamethasone): Patients receive 10mg oral everolimus daily as standard of care and 10ml dexamethasone oral mouthwash, swished for 2-minutes daily, for 8 weeks.
  >>
  >> Dexamethasone: Given as mouthwash
  >>
  >> Questionnaire: Ancillary studies
  >>
  >> Quality-of-Life Assessment: Ancillary studies
  >>
  >> Everolimus: Standard of care
- Group II (Placebo): Patients receive 10mg oral everolimus daily as standard of care and 10ml placebo oral mouthwash, swished for 2-minutes daily, for 8 weeks.
  >>
  >> Placebo: Given as mouthwash
  >>
  >> Questionnaire: Ancillary studies
  >>
  >> Quality-of-Life Assessment: Ancillary studies
  >>
  >> Everolimus: Standard of care
Arm/Group | Group I (Dexamethasone) | Group II (Placebo)
Number analyzed (Participants) | 16 | 17
scores on scale * days | 11.3 (14.83) | 4.6 (6.86)
Statistical Analysis 1: Comparison: Group I (Dexamethasone) vs Group II (Placebo); Test type: Superiority; p = 0.3346, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Incidence of Grade > 2 mIAS as Measured by the SWISH Trial
Description: Original plan for collecting and analyzing this data did not occur due to study termination.
  Grade 2 mIAS is defined as having at least one of the following criteria:>
  1. Oral intake assessed at 50 on the Normalcy of Diet Scale
  2. Patient's reported oral pain (using visual analogue scale 0-10) that meets one of the following: rating of 7 on two consecutive days rating of 8, 9, or 10 on any one day. The incidence of grade 2 mIAS for each treatment arm will be compared by a Chi-square test.
Time Frame: Up to 8 weeks
Population: Original plan for collecting and analyzing this data did not occur due to study termination.
Arm/Group | Group I (Dexamethasone) | Group II (Placebo)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Incidence of Mouth Pain
Description: Original plan for collecting and analyzing this data did not occur due to study termination.
  Will determine if the initiation of dexamethasone at the start of everolimus is associated with the incidence and of mild (score of 1-3), moderate (score of 4-6) and severe (score of 7-10) mouth pain as measured by the NAMPS. Will be assessed by Chi-square tests.
Time Frame: Up to 8 weeks
Population: Original plan for collecting and analyzing this data did not occur due to study termination.
Arm/Group | Group I (Dexamethasone) | Group II (Placebo)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time to Development of Mouth Pain
Description: Original plan for collecting and analyzing this data did not occur due to study termination.
  Will determine if the initiation of dexamethasone at the start of everolimus is associated with the time to development of mild (score of 1-3), moderate (score of 4-6) and severe (score of 7-10) mouth pain as measured by the NAMPS. Will be assessed by Kaplan-Meier and cumulative incidence curves.
Time Frame: Up to 8 weeks
Population: Original plan for collecting and analyzing this data did not occur due to study termination.
Arm/Group | Group I (Dexamethasone) | Group II (Placebo)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Quality of Life Assessed by Linear Analogue Self-Assessment
Description: Original plan for collecting and analyzing this data did not occur due to study termination.
  Will determine if the initiation of dexamethasone at the start of everolimus is associated with quality of life is by comparing numerical analogue scale scores as measured by the Linear Analogue Self-Assessment. The Linear Analogue Self Assessment for quality of life is measured on a 0 to 10 scale, with 0 corresponding to "Quality of life as bad as it can be" and 10 corresponding to "Quality of life as good as it can be." Will be assessed by independent samples t-tests.
Time Frame: Up to 8 weeks
Population: Original plan for collecting and analyzing this data did not occur due to study termination.
Arm/Group | Group I (Dexamethasone) | Group II (Placebo)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Mouth/Throat Sore Level of Activity Interference With Daily Activities
Description: Original plan for collecting and analyzing this data did not occur due to study termination.
  Will determine if the initiation of dexamethasone at the start of everolimus is associated with the level of interference with daily activities as measured by the Patient Reported Outcome (PRO) Common Terminology criteria for Adverse Events (CTCAE) mouth/throat item regarding level of interference with daily activities. The PRO-CTCAE mouth/throat item regarding level of interference with daily activities is measured on a Likert 1-5 scale, with 1 corresponding to "Not at all" and 5 corresponding to "Very much." Will be assessed by independent samples t-tests.
Time Frame: Up to 8 weeks
Population: Original plan for collecting and analyzing this data did not occur due to study termination.
Arm/Group | Group I (Dexamethasone) | Group II (Placebo)
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Sleep Level of Activity Interference With Daily Activities
Description: Original plan for collecting and analyzing this data did not occur due to study termination.
  Will determine if the initiation of dexamethasone at the start of everolimus is associated with the level of interference with daily activities as measured by the PRO-CTCAE sleep item regarding level of interference with daily activities. The PRO-CTCAE sleep item regarding level of interference with daily activities is measured on a Likert 1-5 scale, with 1 corresponding to "Not at all" and 5 corresponding to "Very much." Will be assessed by independent samples t-tests.
Time Frame: Up to 8 weeks
Population: Original plan for collecting and analyzing this data did not occur due to study termination.
Arm/Group | Group I (Dexamethasone) | Group II (Placebo)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Adherence to Everolimus Therapy Dose
Description: Original plan for collecting and analyzing this data did not occur due to study termination.
  Will compare mean daily dose of everolimus between the arms. The mean daily dose of everolimus over 8 weeks will be compared between study arms using independent samples t-tests.
Time Frame: Up to 8 weeks
Population: Original plan for collecting and analyzing this data did not occur due to study termination.
Arm/Group | Group I (Dexamethasone) | Group II (Placebo)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Incidence of Patients Stopping Everolimus Early
Description: Original plan for collecting and analyzing this data did not occur due to study termination.
  Will compare the number of patients who stopped everolimus early between the treatment arms. Will be compared using Chi-squared tests.
Time Frame: Up to 8 weeks
Population: Original plan for collecting and analyzing this data did not occur due to study termination.
Arm/Group | Group I (Dexamethasone) | Group II (Placebo)
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Incidence of Patients Reducing Everolimus Dose
Description: Original plan for collecting and analyzing this data did not occur due to study termination.
  Will compare the number of patients who reduced their everolimus dose between the treatment arms. Will be compared using Chi-squared tests.
Time Frame: Up to 8 weeks
Population: Original plan for collecting and analyzing this data did not occur due to study termination.
Arm/Group | Group I (Dexamethasone) | Group II (Placebo)
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Dexamethasone Prescription Fill Rates
Description: Original plan for collecting and analyzing this data did not occur due to study termination.
  Will compare dexamethasone prescription fill rates between the treatment groups. This will be compared using Chi-squared tests.
Time Frame: Up to 8 weeks
Population: Original plan for collecting and analyzing this data did not occur due to study termination.
Arm/Group | Group I (Dexamethasone) | Group II (Placebo)
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Time to Dexamethasone Prescription Fill
Description: Original plan for collecting and analyzing this data did not occur due to study termination.
  Will compare the time to dexamethasone prescription fill between the treatment groups. This will be compared using Kaplan-Meier and cumulative incidence curves.
Time Frame: Up to 8 weeks
Population: Original plan for collecting and analyzing this data did not occur due to study termination.
Arm/Group | Group I (Dexamethasone) | Group II (Placebo)
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Time to Develop Mouth Sores Per Study Arm Assessed by PRO-CTCAE Mouth/Throat Sore Item Regarding Severity
Description: Original plan for collecting and analyzing this data did not occur due to study termination.
  The time to develop at least mild, moderate, or severe (including "Very severe") mouth sores per study arm as measured by the PRO-CTCAE mouth-throat sore item regarding severity. The PRO-CTCAE mouth-throat sore item regarding severity is measured on a Likert 1-5 scale, with 1 corresponding to "None" and 5 corresponding to "Very severe". Will be assessed by Kaplan-Meier and cumulative incidence curves.
Time Frame: Up to 8 weeks
Population: Original plan for collecting and analyzing this data did not occur due to study termination.
Arm/Group | Group I (Dexamethasone) | Group II (Placebo)
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Mean Degrees of Patient-reported Mouth Sores Per Study Arm Assessed by NAMPS
Description: Original plan for collecting and analyzing this data did not occur due to study termination.
  The mean degrees of patient-reported mouth sores per study arm as measured by the NAMPS will be assessed by independent samples t-tests.
Time Frame: Up to 8 weeks
Population: Original plan for collecting and analyzing this data did not occur due to study termination.
Arm/Group | Group I (Dexamethasone) | Group II (Placebo)
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Median Degree of Patient-reported Mouth Sores Per Study Arm Assessed by NAMPS
Description: Original plan for collecting and analyzing this data did not occur due to study termination.
  The median degrees of patient-reported mouth sores per study arm as measured by the NAMPS will be assessed by independent samples t-tests.
Time Frame: Up to 8 weeks
Population: Original plan for collecting and analyzing this data did not occur due to study termination.
Arm/Group | Group I (Dexamethasone) | Group II (Placebo)
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Proportion of Patients Who Experience Grade 2 Stomatitis
Description: Original plan for collecting and analyzing this data did not occur due to study termination.
  The proportion of patients who experience clinician-reported grade 2 stomatitis (as measured by the CTCAE and performed at 1 and 2 months post-baseline) per study arm will be assessed by Chi-squared tests.
Time Frame: Up to 2 months
Population: Original plan for collecting and analyzing this data did not occur due to study termination.
Arm/Group | Group I (Dexamethasone) | Group II (Placebo)
Number analyzed (Participants) | 0 | 0

18. Other Pre Specified Outcome: Incidence Rate of the mTOR Inhibitor-associated Stomatitis (mIAS)-Related Pain Based on Daily Self-reports Via the Numerical Analogue Scale by Sex
Description: NIH-required analysis. The numerical analogue mouth pain score (NAMPS) is a single item measured on a 0 to 10 scale, with 0 corresponding to "No pain" and 10 corresponding to "Pain as bad as it can be." Will compare the incidence rate of any mouth pain (i.e., any score greater than 0) as assessed by the NAMPS between the prevention versus early treatment approaches using a Chi-square test.
Time Frame: Up to 8 weeks
Population: Population is by Sex. Male and Female population combined equals Overall Number of Participants Analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Dexamethasone) | Group II (Placebo)
Number analyzed (Participants) | 16 | 17
Participants
  Female: number analyzed (Participants) | 12 | 15
  Female: No Pain | 5 | 8
  Female: Pain | 7 | 7
  Male: number analyzed (Participants) | 4 | 2
  Male: No Pain | 2 | 0
  Male: Pain | 2 | 2
Statistical Analysis 1: Comparison: Group I (Dexamethasone) vs Group II (Placebo); Female Population; Test type: Superiority; p < 0.70361, Fisher Exact
Statistical Analysis 2: Comparison: Group I (Dexamethasone) vs Group II (Placebo); Male population; Test type: Superiority; p < 0.4667, Fisher Exact

19. Other Pre Specified Outcome: Incidence Rate of the mTOR Inhibitor-associated Stomatitis (mIAS)-Related Pain Based on Daily Self-reports Via the Numerical Analogue Scale by Race
Description: as for outcome 18
Time Frame: Up to 8 weeks
Population: Black or African American population is different than white population
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Dexamethasone) | Group II (Placebo)
Number analyzed (Participants) | 16 | 17
Participants
  Black or African American: number analyzed (Participants) | 4 | 1
  Black or African American: No Pain | 1 | 0
  Black or African American: Pain | 3 | 1
  White: number analyzed (Participants) | 12 | 16
  White: No Pain | 6 | 8
  White: Pain | 6 | 8
Statistical Analysis 1: Comparison: Group I (Dexamethasone) vs Group II (Placebo); Black or African American population; Test type: Superiority; p < 1.0, Fisher Exact
Statistical Analysis 2: Comparison: Group I (Dexamethasone) vs Group II (Placebo); White population; Test type: Superiority; p < 1.0, Fisher Exact

20. Other Pre Specified Outcome: Incidence Rate of the mTOR Inhibitor-associated Stomatitis (mIAS)-Related Pain Based on Daily Self-reports Via the Numerical Analogue Scale by Ethnicity.
Description: as for outcome 18
Time Frame: Up to 8 weeks
Population: Population is by Ethnicity. Not Hispanic or Latino and Other population combined equals Overall Number of Participants Analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Dexamethasone) | Group II (Placebo)
Number analyzed (Participants) | 16 | 17
Participants
  Not Hispanic or Latino: number analyzed (Participants) | 15 | 16
  Not Hispanic or Latino: No Pain | 6 | 7
  Not Hispanic or Latino: Pain | 9 | 9
  Other: number analyzed (Participants) | 1 | 1
  Other: No Pain | 1 | 1
  Other: Pain | 0 | 0
Statistical Analysis 1: Comparison: Group I (Dexamethasone) vs Group II (Placebo); Not Hispanic or Latino population; Test type: Superiority; p < 1.0, Fisher Exact

21. Other Pre Specified Outcome: Severity of Mouth Pain Scores by Sex
Description: as for outcome 2
Time Frame: Up to 8 weeks
Population: Population is by Sex. Male and Female population combined equals Overall Number of Participants Analyzed.
Measure: Mean (Inter-Quartile Range); unit: scores on scale * days
Arm/Group | Group I (Dexamethasone) | Group II (Placebo)
Number analyzed (Participants) | 16 | 17
scores on scale * days
  Female: number analyzed (Participants) | 12 | 15
  Female | 11.4 [0.0 to 47.3] | 2.7 [0.0 to 15.7]
  Male: number analyzed (Participants) | 4 | 2
  Male | 11.0 [0.0 to 33.4] | 18.8 [17.0 to 20.7]
Statistical Analysis 1: Comparison: Group I (Dexamethasone) vs Group II (Placebo); Female population; Test type: Superiority; p < 0.1701, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group I (Dexamethasone) vs Group II (Placebo); Male population; Test type: Superiority; p < 0.4811, Wilcoxon (Mann-Whitney)

22. Other Pre Specified Outcome: Severity of Mouth Pain Scores by Race
Description: as for outcome 2
Time Frame: Up to 8 weeks
Population: Population is by Race. Black or African American and White population combined equals Overall Number of Participants Analyzed.
Measure: Mean (Inter-Quartile Range); unit: scores on scale * days
Arm/Group | Group I (Dexamethasone) | Group II (Placebo)
Number analyzed (Participants) | 16 | 17
scores on scale * days
  Black or African American: number analyzed (Participants) | 4 | 1
  Black or African American | 9.3 [0.0 to 22.8] | 7.9 [7.9 to 7.9]
  White: number analyzed (Participants) | 12 | 16
  White | 12.0 [0.0 to 47.3] | 4.4 [0.0 to 20.7]
Statistical Analysis 1: Comparison: Group I (Dexamethasone) vs Group II (Placebo); Black or African American Population; Test type: Superiority; p < 1.0, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group I (Dexamethasone) vs Group II (Placebo); White Population; Test type: Superiority; p < 0.5029, Wilcoxon (Mann-Whitney)

23. Other Pre Specified Outcome: Severity of Mouth Pain Scores by Ethnicity
Description: as for outcome 2
Time Frame: Up to 8 weeks
Population: as for outcome 20
Measure: Mean (Inter-Quartile Range); unit: scores on scale * days
Arm/Group | Group I (Dexamethasone) | Group II (Placebo)
Number analyzed (Participants) | 16 | 17
scores on scale * days
  Not Hispanic or Latino: number analyzed (Participants) | 15 | 16
  Not Hispanic or Latino | 12.1 [0.0 to 47.3] | 4.9 [0.0 to 20.7]
  Other: number analyzed (Participants) | 1 | 1
  Other | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
Statistical Analysis 1: Comparison: Group I (Dexamethasone) vs Group II (Placebo); Not Hispanic or Latino Population; Test type: Superiority; p < 0.2950, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: 3 patients in Dexamethasone Arm withdrew prior to starting treatment and no AE data was collected. Out of 20 randomized patients in Dexamethasone arm, 17 patients had AE data. 1 patient in Placebo Arm had a protocol violation. Patient did no start Everolimus and no AE data was collected. Out of 19 randomized patients in Placebo arm, 18 patients had AE data.
Arm/Group | Group II (Placebo) | Group I (Dexamethasone)
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 3/18 | 2/17
Other Adverse Events (participants affected / at risk) | 16/18 | 12/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group II (Placebo) (N=18) | Group I (Dexamethasone) (N=17)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group II (Placebo) (N=18) | Group I (Dexamethasone) (N=17)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 2 (5) | 0 (0)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 6 (15) | 7 (29)
Nausea (Gastrointestinal disorders) | 3 (6) | 2 (2)
Oral pain (Gastrointestinal disorders) | 6 (16) | 7 (29)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 14 (57) | 9 (36)
Mucosal infection (Infections and infestations) | 0 (0) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (3) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (4) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (14) | 6 (15)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Dysgeusia (Nervous system disorders) | 2 (5) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 9 (40) | 4 (20)
Irritability (Psychiatric disorders) | 3 (10) | 2 (4)
Breast pain (Reproductive system and breast disorders) | 1 (3) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (4) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-14): https://cdn.clinicaltrials.gov/large-docs/40/NCT03839940/Prot_SAP_000.pdf